CLINICAL TRIAL: NCT03700957
Title: A Clinical Study on the Impact of Docosahexaenoic Acid on the Prevention of Necrotizing Enterocolitis in Preterm Neonates
Brief Title: The Impact of Docosahexaenoic Acid on the Prevention of Necrotizing Enterocolitis in Preterm Neonates
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Ain Shams University (Other)
Responsible Party: Principal Investigator, Dina Khaled Mohamed Abou El Fadl, Assistant Lecturer, Future University in Egypt
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 73
Record Dates: First submitted 2018-09-29; First posted 2018-10-09 (Actual); Last update posted 2018-10-09 (Actual); Status verified 2018-10

CONDITIONS: Necrotizing Enterocolitis
MeSH Terms: conditions — Enterocolitis, Necrotizing | interventions — Docosahexaenoic Acids

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Docosahexaenoic Acid Group (Experimental): participants will recieve 100 milligrams of Docosahexaenoic Acid per day for 14 days
  Interventions: Dietary Supplement: Docosahexaenoic Acid
- Control Group (Placebo Comparator): participants will recieve placebo
  Interventions: Other: placebo

INTERVENTIONS:
Dietary Supplement: Docosahexaenoic Acid — 100 milligrams of Docosahexaenoic Acid
  Arms: Docosahexaenoic Acid Group
Other: placebo — placebo
  Arms: Control Group

SUMMARY:
The study will assess the efficacy of Docosahexaenoic Acid in reducing the incidence of necrotizing enterocolitis in premature infants.

DETAILED DESCRIPTION:
The efficacy of Docosahexaenoic Acid in reducing the incidence of necrotizing enterocolitis in preterm neonates will be evalutaed through measuring its immune-modulatory effect on proinflammatory cytokines.

ELIGIBILITY:
Inclusion Criteria:

* Preterm neonates having a gestational age equal or less than 34 weeks at birth.
* Weight (less than or equal 1.500 KG)
* Clinically stable to begin enteral feeding

Exclusion Criteria:

* Persistent bleeding at any level.
* Receiving medication to avoid coagulation.
* Persistent vomiting.
* Gastrointestinal malformations.
* Mother taking Omega-3 supplements and planning to breastfeed.

Ages: 1 Day to 3 Weeks | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 60 (Estimated)
Dates: Start 2018-10 (Estimated); Primary Completion 2019-06 (Estimated); Study Completion 2019-09 (Estimated)

PRIMARY OUTCOMES:
Efficacy of Docosahexaenoic Acid in reducing the incidence of Necrotizing Enterocolitis in premature infants. | 10 days
  Monitoring the change in the serum levels of Interleukin-1 beta

CONTACTS AND LOCATIONS:
Overall Officials: Dina Abou El Fadl, Msc., Principal Investigator — Future University in Egypt

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Shulhan J, Dicken B, Hartling L, Larsen BM. Current Knowledge of Necrotizing Enterocolitis in Preterm Infants and the Impact of Different Types of Enteral Nutrition Products. Adv Nutr. 2017 Jan 17;8(1):80-91. doi: 10.3945/an.116.013193. Print 2017 Jan. PMID 28096129
- [Background] Baack ML, Puumala SE, Messier SE, Pritchett DK, Harris WS. Daily Enteral DHA Supplementation Alleviates Deficiency in Premature Infants. Lipids. 2016 Apr;51(4):423-33. doi: 10.1007/s11745-016-4130-4. Epub 2016 Feb 4. PMID 26846324
- [Derived] Abou El Fadl DK, Ahmed MA, Aly YA, Darweesh EAG, Sabri NA. Impact of Docosahexaenoic acid supplementation on proinflammatory cytokines release and the development of Necrotizing enterocolitis in preterm Neonates: A randomized controlled study. Saudi Pharm J. 2021 Nov;29(11):1314-1322. doi: 10.1016/j.jsps.2021.09.012. Epub 2021 Sep 25. PMID 34819793